CLINICAL TRIAL: NCT05865015
Title: Dietary Patterns, Physical Activity Level, Body Composition and Serum Vitamin B9, Vitamin B12 and Vitamin D Levels in Women Undergoing in Vitro Fertilization and the Outcomes of in Vitro Fertilization
Brief Title: Nutritional Status of Women Undergoing in Vitro Fertilization
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor
Other Study IDs: TP20210218
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-02

CONDITIONS: IVF; Body Weight; Nutrient Deficiency; Dietary Vitamin B12 Deficiency Anemia; Dietary Folate Deficiency Anemia
Keywords: Dietary Patterns; Mediterranean diet; In Vitro Fertilization; Diet; Fertility; Infertility; Assisted Reproduction
MeSH Terms: conditions — Body Weight; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — The patient will have blood drawn for biochemical laboratory tests at the Clinical Institute of Clinical Chemistry and Biochemistry, University Clinical Centre Ljubljana (in addition to the standard tests, the investigators will also determine vitamin B9 or folate and folic acid, vitamin B12, vitamin D, oligoelements, heavy metals, hormone disruptors, etc.) The protection of personal data will be guaranteed, as each blood sample will be labelled or recorded during the study under a code identical to the code of the questionnaire completed by the patient. Information on the results of the IVF/ICSI procedure will be obtained from the patients' medical records with their consent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:

SUMMARY:
Infertility affects around 15 % of couples in their reproductive years. Even though the use of assisted reproductive technologies (ART) in aforementioned couples is increasing, their success rate is still relatively low. Hence it is important to identify and better understand potential modifiable dietary and lifestyle risk factors that may influence the success of ART. This study will include women undergoing IVF with a view to investigating the relationship between preconception dietary patterns, body composition, physical activity level, serum values of vitamin B9, vitamin B12 and vitamin D and the outcomes of IVF, such as the number of obtained oocytes, fertilization rate and clinical pregnancy. Main hypothesis is that women undergoing IVF, who eat a balanced diet, maintain healthy body weight and have adequate serum levels of vitamin B9, vitamin B12 and vitamin D, have a higher chance of achieving better IVF outcomes.

DETAILED DESCRIPTION:
Infertility, which affects around 15 % of couples of reproductive, refers to the inability of a couple to conceive after 12 months of unprotected sex. Pre-conception dietary habits have been shown to influence the outcomes of the in vitro fertilization (IVF) procedure, such as oocyte and embryo quality, embryo implantation and successful pregnancy. Thus far, a balanced diet, especially a Mediterranean diet (MED), is known to have a beneficial effect on the outcome of IVF in women before the IVF process. MED is characterised by a high intake of antioxidants that reduces oxidative stress, which otherwise increases the likelihood of infertility in women. In addition, the Mediterranean diet is characterised by a higher intake of folate and polyunsaturated omega-3 fatty acids (especially eicosapentaenoic acid), which also has a beneficial effect on the outcome of the IVF process. While some authors have not confirmed that the Mediterranean diet can increase the likelihood of pregnancy after IVF in infertile women, they have found that it can increase the number of embryos ready for transfer. On the other hand, an unbalanced diet with a typically low intake of vitamins and minerals has an adverse effect on fertility. Low intakes of vitamins B6, B9 and B12 are particularly problematic, as their deficiency leads to the accumulation of homocysteine, which can lead to hyperhomocysteinemia. Elevated levels of homocysteine in follicular fluid are known to negatively affect the number of retrieved oocytes and embryo quality in IVF and intracytoplasmic sperm injection (ICSI). Higher serum levels of vitamin B9 and vitamin B12 in women have been shown to increase the likelihood of a live birth after ART, as they have a beneficial effect on pregnancy maintenance after embryo implantation. Despite the known importance of sufficient vitamin B9 and vitamin B12 intake to support fertility and success of the IVF procedure, some women undergoing IVF still have largely insufficient serum levels of vitamin B9 and vitamin B12 prior to the IVF procedure. Vitamin D deficiency in women has also been identified as a modifiable risk factor that may affect the outcome of ART. Vitamin D is involved in steroid formation in the ovary and in the expression of genes in the endometrium that are crucial for embryo implantation. For this reason, women should have their serum vitamin D levels routinely checked before IVF. This would allow women with an identified vitamin D deficiency to start vitamin D supplementation, which may have a beneficial effect on IVF outcome. Another modifiable factor with an impact on ART outcome is excessive body weight and obesity, as adipose tissue interferes with the synthesis and bioavailability of sex hormones in women, which negatively affects oocyte quality and endometrial receptivity. In this group of women, oocytes are less likely to properly develop after IVF than oocytes from women with optimal body weight. In addition, it is known that women who are overweight or obese have a lower probability of embryo implantation, clinical pregnancy and live birth after IVF/ICSI. However, in women with obesity, regular physical activity can have a positive effect on IVF/ICSI outcomes even when body mass index is unchanged. Consequently, the time before the ART procedure presents an opportunity to establish nutritional counselling to facilitate women's achievement of optimal body weight and intake of the necessary micronutrients, which could positively influence the outcome of the ART procedure. However further studies on the impact of women's dietary habits and nutritional status on the outcome of the ART procedure are urgently needed before this can be done.

The investigators aim to identify which modifiable risk factors for IVF/ICSI failure are poorly managed in women and to improve understanding of the impact of women's dietary habits, physical. The investigators are interested in whether women have a balanced diet before the IVF/ICSI procedure and whether they successfully prevent vitamin B9, vitamin B12 and vitamin D deficiencies, which can negatively affects the outcomes of IVF/ICSI. By measuring women's body composition before IVF/ICSI, the investigators aim to test whether an excessive percentage of fat mass reduces the likelihood of IVF/ICSI success, as suggested by the scientific evidence to date. The information obtained will allow the design of future nutritional counselling for women before IVF/ICSI to facilitate the establishment of a healthier lifestyle and potentially increase the likelihood of success of the IVF/ICSI procedure, thereby reducing the economic burden of infertility treatment. In the first study of its kind in Slovenia, the investigators expect to identify the association between dietary habits, physical activity levels, body composition and serum levels of vitamin B9, vitamin B12 and vitamin D and IVF/ICSI outcomes, such as the number of retrieved oocytes, the rate of fertilisation of oocytes and clinical pregnancy, in women prior to undergoing IVF/ICSI. The underlying hypothesis is that women who have a balanced diet and lead a healthier lifestyle prior to IVF/ICSI will have a higher likelihood of favourable IVF/ICSI outcomes.

The research will be conducted at the Clinical Department of Reproduction, Department of Gynaecology, University Clinical Centre Ljubljana, with the collaboration of the Faculty of Biotechnology, University of Ljubljana. The study will be cross-sectional, non-interventional. Patients will be introduced to the study and its process at the time of entering the IVF/ICSI procedure. If the patient signs the informed consent form, the investigators will obtain her height and weight measurement and body composition measurement by non-invasive bioimpedance analysis. The patient will also fill in the questionnaire required for the study, which includes questions regarding sociodemographic status, dietary habits, frequency of food consumption in the past month, and physical activity level. In addition, prior to the IVF/ICSI procedure, the patient will have blood drawn for biochemical laboratory tests at the Clinical Institute of Clinical Chemistry and Biochemistry, University Clinical Centre Ljubljana (in addition to the standard tests, the investigators will also determine vitamin B9 or folate and folic acid, vitamin B12, vitamin D, oligoelements, heavy metals, hormone disruptors, etc.) The protection of personal data will be guaranteed, as each blood sample will be labelled or recorded during the study under a code identical to the code of the questionnaire completed by the patient. Information on the results of the IVF/ICSI procedure will be obtained from the patients' medical records with their consent. Statistical evaluation of the data will be performed at the Faculty of Biotechnology, University of Ljubljana. The data obtained will be subjected to appropriate statistical analysis to determine the association of dietary habits, body composition, physical activity level and serum vitamin B9, vitamin B12 and vitamin D levels of patients before the IVF/ICS procedure on IVF/ICS outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing IVF/ICSI treatment

Exclusion Criteria:

* Women's age > 39
* Endometriosis

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women undergoing IVF treatment at the University Medical Centre Ljubljana.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-09-10 (Actual)

PRIMARY OUTCOMES:
Oocyte number | 3 months
  Total Number of oocytes produced.

SECONDARY OUTCOMES:
Fertilization rate | 3 months
  Fertilization rate will be determined on day 1 after the IVF/intracytoplasmatic sperm injection procedure, and is going to calculated as the number of fertilized oocytes divided by the total number of oocytes retrieved.

OTHER OUTCOMES:
Clinical pregnancy rate | 6 months
  Elevation in b-human chorionic gonadotropin with the confirmation of an intrauterine pregnancy by ultrasound, first performed at 6 weeks of gestation

CONTACTS AND LOCATIONS:
Locations (2):
- Slovenia (2):
  - Division of Ob/Gyn, University Medical Centre Ljubljana, Ljubljana
  - Division of Peadiatrics, University Medical Centre Ljubljana, Ljubljana

IPD SHARING:
Plan to Share IPD: Undecided